CLINICAL TRIAL: NCT06335563
Title: Application of Intelligent Augmented Reality Glasses in Assisting the Localization of Small Pulmonary Nodules:A Prospective, Randomized, Controlled, Noninferiority Trial
Brief Title: Augmented Reality Navigation Versus Traditional CT Guidance for Preoperative Localization of Pulmonary Nodules
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Deping Zhao, Administrative Director of Thoracic Surgery Department, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STAR009
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Pulmonary Nodule

STUDY DESIGN:
Intervention Model Description: AR glasses-assisted puncture localizing group versus CT-guided conventional pulmonary nodule puncture localizing group
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AR glasses-assisted pulmonary nodule puncture localization (Experimental): Combined with placing positioning marks on the patient's body surface and tracing the needle entry point with the assistance of a CT scan gantry laser. Disinfect the area around the puncture needle point, and use 2% lidocaine for local infiltration anesthesia. The doctor wears augmented reality (AR) glasses, completes the connection between the AR glasses and the puncture target, and clicks on the puncture point plane through the puncture target needle tip. Calibrate the puncture position at any two points. After confirming that the patient has held his breath, quickly puncture the needle into the pleura and advance it to the planned puncture position according to the screen prompts. After the second CT scan is performed to confirm that the puncture needle is positioned at a reasonable position, the positioning hook wire is released and the puncture needle sheath is withdrawn.
  Interventions: Procedure: AR glasses-assisted pulmonary nodule puncture localization
- CT-guided pulmonary nodule puncture localization (Active Comparator): Positioning markers are placed on the patient's surface and the first CT scan is performed. The needle insertion point and needle insertion depth are designed based on the two-dimensional CT scan image and the positioning marks. The location of the needle entry point was traced with the laser assistance of the CT gantry. Disinfect and puncture around the needle point, and use 2% lidocaine for local infiltration anesthesia. According to the designed needle path angle, the needle is first inserted under the skin, and a second CT scan is performed to confirm that the extension line of the puncture needle is within the nodule range. Then the needle is inserted to the target depth, and the third CT scan is performed. After confirming that the puncture needle is positioned at a reasonable position, the positioning hook wire is released and the puncture needle sheath is withdrawn.
  Interventions: Procedure: CT-guided pulmonary nodule puncture localization

INTERVENTIONS:
Procedure: AR glasses-assisted pulmonary nodule puncture localization — Combined with placing positioning marks on the patient's body surface and tracing the needle entry point with the assistance of a CT scan gantry laser. Disinfect the area around the puncture needle point, and use 2% lidocaine for local infiltration anesthesia. The doctor wears augmented reality (AR) glasses, completes the connection between the AR glasses and the puncture target, and clicks on the puncture point plane through the puncture target needle tip. Calibrate the puncture position at any two points. After confirming that the patient has held his breath, quickly puncture the needle into the pleura and advance it to the planned puncture position according to the screen prompts. After the second CT scan is performed to confirm that the puncture needle is positioned at a reasonable position, the positioning hook wire is released and the puncture needle sheath is withdrawn.
  Arms: AR glasses-assisted pulmonary nodule puncture localization
Procedure: CT-guided pulmonary nodule puncture localization — Positioning markers are placed on the patient's surface and the first CT scan is performed. The needle insertion point and needle insertion depth are designed based on the two-dimensional CT scan image and the positioning marks. The location of the needle entry point was traced with the laser assistance of the CT gantry. Disinfect and puncture around the needle point, and use 2% lidocaine for local infiltration anesthesia. According to the designed needle path angle, the needle is first inserted under the skin, and a second CT scan is performed to confirm that the extension line of the puncture needle is within the nodule range. Then the needle is inserted to the target depth, and the third CT scan is performed. After confirming that the puncture needle is positioned at a reasonable position, the positioning hook wire is released and the puncture needle sheath is withdrawn.
  Arms: CT-guided pulmonary nodule puncture localization

SUMMARY:
This study aims to conduct a large-sample randomized controlled clinical trial, using traditional CT-guided thoracic puncture localization as a comparison, to explore the accuracy, safety and clinical advantages of Intelligent AR glasses in assisting preoperative localizing of small pulmonary nodules.

DETAILED DESCRIPTION:
This study is an open-label prospective single-center non-inferiority randomized controlled clinical trial. Patients in the Pulmonary Hospital Affiliated to Tongji University who are scheduled to undergo percutaneous puncture localization of small pulmonary nodules are used as the research subjects. According to the entry and exit criteria Patients were included in the clinical trial, and the enrolled patients were randomly divided into the AR glasses-assisted puncture localizing group (experimental group) and the CT-guided conventional pulmonary nodule puncture localizing group (control group), aiming to evaluate the puncture of pulmonary nodules guided by Intelligent AR glasses. Non-inferiority of localization compared with conventional CT-guided pulmonary nodule puncture localization.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80, no gender limit;
2. Chest CT shows that the nodule involves the outer third of the lung and can be removed by wedge resection;
3. Chest CT (lung window mode), the maximum diameter of the nodule is ≤2 cm;
4. Physical condition score ECOG 0-2 points;
5. If you plan to undergo percutaneous puncture and localization of small pulmonary nodules, the puncture needle path will be determined by the attending physician;
6. Patients voluntarily participate and sign informed consent.

Exclusion Criteria:

1. The lesion is located in front of the scapula, and the needle path is blocked;
2. The distance between the center of the lesion and the top of the diaphragm is < 3 cm;
3. The lesion is adjacent to the hilus or large blood vessels;
4. Pleural adhesions caused by a history of thoracotomy or pleural infection;
5. The patient voluntarily withdraws midway.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of puncture localization of pulmonary nodules | Intraoperative
  Quantified as the shortest distance from the actual position of the puncture needle tip to the originally planned puncture point

SECONDARY OUTCOMES:
Success rate of puncture localization of pulmonary nodules | Intraoperative
  The puncture is defined as successful when the distance between the actual localizing point of the puncture needle tip and the center of the localized nodule does not exceed 20 mm.
Adjust the number of needle punctures | Intraoperative
  Number of needle insertion attempts required for successful localizing
Operating time | Intraoperative
  The time span from the patient's first CT scan to the last CT scan, in minutes
Radiation dose | Intraoperative
  The length product value of the radiation dose recorded by the CT scanner, measured in mGy * cm

CONTACTS AND LOCATIONS:
Overall Officials: Deping Zhao, MD, PhD, Principal Investigator — Shanghai Pulmonary Hospital, School of Medicine, Tongji University
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China